CLINICAL TRIAL: NCT06508242
Title: Effects Of Vitamin D On Bone, Muscle, And Adipose Tissue In Obese Subjects: A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Effects Of Vitamin D On Bone, Muscle, And Adipose Tissue In Obese Subjects
Acronym: DON3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 73.20
Record Dates: First submitted 2024-03-25; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-03

CONDITIONS: Musculoskeletal Diseases; Inflammation; Sarcopenic Obesity
MeSH Terms: conditions — Musculoskeletal Diseases; Inflammation | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D intervention group (Active Comparator): 50.000 IU of oral cholecalciferol/week
  Interventions: Drug: Cholecalciferol
- Placebo group (Placebo Comparator): Placebo treatment/week
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — cholecalciferol
  Arms: Vitamin D intervention group
Other: Placebo — placebo
  Arms: Placebo group

SUMMARY:
Obesity has emerged as a risk factor in the onset of bone, muscle and adipose tissue impairments that are further aggravated by vitamin D deficiency. A link of an active bone-muscle-adipose axis is represented by Wnt pathway. This study will test the hypothesis that vitamin D improves bone, muscle, and adipose tissue health through a positive modulation of Wnt pathway. It will be carried out a double-blind, placebo-controlled study of cholecalciferol supplementation in vitamin D-deficient obese adults. Specific aims will be: 1) to test the direct effect of vitamin D on Wnt signaling in bone, muscle, and adipose tissue; 2) to evaluate muscle mass and strength; 3) to assess changes in vitamin D status across different administration strategy (weekly, fortnightly, monthly).

This study will provide not only insight of new mechanisms involved in the pathophysiology of obesity-related musculoskeletal impairments but also evidence for new treatment recommendations for vitamin D deficiency in obesity.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory willing and able to provide informed consent;
* post-menopausal women (55-75 y.o.) and age-matched men;
* BMI 30 >= kg/m2;
* serum 25OHD < 20 ng/ml
* hip replacement surgery due to osteoarthritis according to orthopedic clinical decision

Exclusion Criteria:

* eGFR <40 ml/min/1.72 m2 by EPI formula (21);
* hypercalcemia (>10.5 mg/dL);
* osteoporosis (hip or vertebral t-score >-2.5);
* conditions affecting bone
* vitamin D and/or calcium metabolism (chronic liver disease, renal failure, malabsorption, hypercortisolism);
* medications altering bone metabolism (e.g. denosumab, bisphosphonates, teriparatide, glucocorticoids, aromatase inhibitors, estrogen);
* enrollment in an interventional clinical trial in the previous 3 months.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
WNT pathway regulation | from 6 to 30 months
  Specifically, WNT10b, WNT5a, sFRP5, pGSK-3ß-Ser9 and total GSK-3ß expression will be evaluated and subsequently confirmed by RT-PCR and Western-blot analysis on adipose and muscle tissue. Serum sclerostin,DDK-1 and sFRP5 will be also evaluated by ELISA

SECONDARY OUTCOMES:
Muscle strength and function | from 0 to 32 months
  • Gene involved in myogenesis will be analyzed by RT-PCR (Relative Expression) and Western-blot (Relative Abundance).
Muscle strength and function | from 0 to 32 months
  • RNAseq will be performed on muscle biopsies to address changes in the transcript profile and subsequent gene enrichment analysis related to vitamin D supplementation
Muscle strength and function | from 0 to 32 months
  • Exosomal-miRNAs will be isolated from treated and untreated adipose tissue with Vitamin D
Muscle strength and function | from 0 to 32 months
  Following tests will be performed:
  • MRI and total body DXA to characterize muscle health status and muscle quality
Muscle strength and function | from 0 to 32 months
  • Muscle quality will be assessed also by calculating the ratio of Lower extremity (LE) strength to LE lean body mass (by DXA, g/cm^2)
Muscle strength and function | from 0 to 32 months
  • Handled dynamometer (to test muscle strength, Kg).
Muscle strength and function | from 0 to 32 months
  • Physical performance evaluation by modified and gait-speed test (m/s).
Muscle strength and function | from 0 to 32 months
  • Validated questionnaires for sarcopenia assessment such as SARC-F and MSRA (Units on a scale)
Effects of inflammation and WNT pathway on adipose tissue | from 0 to 32 months
  • Analysis of gene and protein expression of molecules related to Inflammation and the effects of WNT pathway on adipose tissue
Effects of inflammation and WNT pathway on adipose tissue | from 0 to 32 months
  • RNA transcription will be performed as described above, as well as exosome analysis.
Effects of inflammation and WNT pathway on bone tissue | from 0 to 32 months
  • Analysis of gene expression of the genes related to WNT pathway
Effects of inflammation and WNT pathway on bone tissue | from 0 to 32 months
  • An immunohistochemistry assay will be performed on the bone to analyze the number and localisation of Teff and Treg cells.
Effects of inflammation and WNT pathway on bone tissue | from 0 to 32 months
  • Synovial fluid: measurement of pro- and anti-inflammatory/metabolic molecules using the Luminex technology

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico di Roma, Roma, RM, Italy